CLINICAL TRIAL: NCT02346422
Title: A Phase 1/2 Study of the Safety and Preliminary Activity of MYDICAR® at a Dose of 2.5 x 10^13 DNase Resistant Particles (DRP) in Subjects With Advanced Heart Failure Divided Into 2 Phases: Phase 1 Open-label and Phase 2 Randomized, Double-blind, Placebo-controlled
Brief Title: A Phase 1/2 Study of High-dose Genetically Targeted Enzyme Replacement Therapy for Advanced Heart Failure
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor has suspended clinical development of MYDICAR for heart failure.
Sponsor: Celladon Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CELL-009
Record Dates: First submitted 2015-01-15; First posted 2015-01-27 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Ischemic Cardiomyopathy; Non-ischemic Cardiomyopathy; Heart Failure; Cardiomyopathies
Keywords: Heart Failure; Cardiomyopathies; Heart Diseases; Cardiovascular Diseases; Cardiomegaly; Gene Therapy
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Heart Diseases; Cardiovascular Diseases; Cardiomegaly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MYDICAR (Experimental): Single intracoronary infusion of MYDICAR, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 2.5 x 10^13 DRP. Administered in MYDICAR Phase 1 and MYDICAR Phase 2.
  Interventions: Genetic: MYDICAR Phase 1; Genetic: MYDICAR Phase 2
- Placebo (Placebo Comparator): Single intracoronary infusion of placebo (Sodium Chloride Injection, USP) (Placebo Phase 2 only).
  Interventions: Genetic: Placebo Phase 2 only

INTERVENTIONS:
Genetic: MYDICAR Phase 1 — Single dose of MYDICAR
  Other Names: AAV1/SERCA2a
  Arms: MYDICAR
Genetic: MYDICAR Phase 2 — Single dose of MYDICAR
  Other Names: AAV1/SERCA2a
  Arms: MYDICAR
Genetic: Placebo Phase 2 only — Single dose of placebo
  Arms: Placebo

SUMMARY:
The purpose of this trial is to characterize the safety profile and preliminary activity of high-dose MYDICAR® in persons with advanced heart failure when added to their maximal and optimized therapy.

DETAILED DESCRIPTION:
Heart failure (HF) is a disabling chronic disease and the most frequent discharge diagnosis for hospitalization among older adults.The American Heart Association (AHA) 2006 update on heart disease reported that 5 million Americans are believed to have symptomatic HF, and 550,000 patients are newly diagnosed each year. The estimated direct and indirect cost of HF in the United States (U.S.) for 2006 was ~$29.6 billion. Despite the significant resources expended on the treatment of this disease, outcomes remain poor. The five-year survival for individuals diagnosed with HF is less than 50%, and in end-stage HF, the one-year survival may be as low as 25% regardless of medical therapy.

Recent studies suggest that the failing heart is not refractory to treatment, as was previously believed. For example, the observation that a small percentage of subjects with left ventricular assist devices can be permanently weaned from their device strongly suggests that damaged hearts are capable of recovering lost function.

Celladon Corporation (Celladon) is investigating gene transfer as a method to restore calcium ion (Ca++) cycling in HF patients. The gene therapy vehicle uses a recombinant adeno-associated viral vector (AAV), which consists of an AAV serotype 1 capsid and contains the human sarcoplasmic reticulum Ca++ ATPAse (SERCA2a) complementary DNA (cDNA) flanked by inverted terminal repeats derived from AAV serotype 2 (AAV1/SERCA2a). MYDICAR® refers to AAV1/SERCA2a drug product intended for administration by percutaneous delivery. Phase 1/2 clinical trials have demonstrated initial safety and evidence of improvement in clinical outcomes at MYDICAR doses of up to 1 x 10^13 DNase-resistant particles (DRP). The trial described here is designed to investigate the safety profile and preliminary activity of MYDICAR at a dose of 2.5 x 10^13 DRP; this dose is 2.5-fold higher than previously investigated doses.

ELIGIBILITY:
Inclusion Criteria:

* Unless otherwise specified, screening must be performed within 30 days prior to enrollment (phase 1) or enrollment/randomization (phase 2) except as noted below. Subjects must meet the following criteria to be eligible for the study:

  1. AAV1 neutralizing antibodies (NAb) negative (titer <1:2 or equivocal) within 60 days prior to screening.
  2. Age 18-80 years, inclusive, at the time of signing the first informed consent.
  3. Chronic ischemic or non-ischemic cardiomyopathy, except for hypertrophic cardiomyopathy. Toxic or alcoholic cardiomyopathies are allowed as long as toxin or alcohol exposure has been eliminated and a sufficient amount of time has elapsed to rule out spontaneous recovery. Similarly, patients with viral or peripartum cardiomyopathy will not be enrolled until sufficient time has elapsed to rule out spontaneous recovery. Subjects with ischemic cardiomyopathy must have at least 1 major coronary vessel with thrombolysis in myocardial infarction (TIMI) grade 3 flow. (If a subject has not undergone recent coronary angiography, TIMI flow may be assessed during the study angiography just prior to investigational medicinal product [IMP] infusion).
  4. Left ventricular ejection fraction ≤35%.
  5. Diagnosis of New York Heart Association class III/IV heart failure (HF) for a minimum of 60 days prior to screening.
  6. For phase 2 only, the presence of at least one of the following risk factors:

     1. Hospitalization for HF within 6 months of screening, or in lieu of hospitalization, at least 2 outpatient interventions for the intended treatment of signs and symptoms of worsening HF (e.g., intravenous [IV] diuretics, peripheral ultrafiltration).
     2. N-terminal prohormone brain natriuretic peptide (NT-proBNP) >1200 pg/mL within 30 days of screening; if subject is in atrial fibrillation, NT-proBNP >1600 pg/mL within 30 days of screening.
  7. Individualized, maximal, optimized HF therapy consistent with American College of Cardiology/American Heart Association practice guidelines for the treatment of chronic heart failure (ACC/AHA HF guidelines) and as updated from time to time:

     1. Medical therapy, as appropriate to the individual subject, including oral diuretic, angiotensin-converting enzyme (ACE) inhibitor or, if ACE intolerant, angiotensin-receptor blocker and beta blocker at approved dosages as labeled in the respective package insert and optimized for the subject.

        * The choice of beta blocker is limited to those approved for HF (bisoprolol, carvedilol or metoprolol succinate). Metoprolol tartrate is not approved for HF and is not allowed.
        * Unless contraindicated or not tolerated, the addition of an aldosterone antagonist should be considered in the absence of hyperkalemia and significant renal dysfunction and according to evolving standards. However, the final decision is at the discretion of the investigator.
        * Dosing of the above medications must be stable for a minimum of 30 days prior to screening, although up- or down-titration of diuretics, as medically indicated, is permitted.
        * Patients requiring IV diuretics during this period will be required to undergo an additional 30 day period of stabilization on oral diuretics.
        * Enrollment of any subject with any deviation from these criteria must be preapproved by the medical monitor.
     2. Resynchronization therapy, if clinically indicated according to ACC/AHA HF guidelines, must have been initiated at least 6 months prior to screening.
     3. If the subject is already participating in a cardiac rehabilitation program, it should be consistent with the current clinical practice and guidelines and continue at least through the 12-Month Active Observation Period. This does not imply that the potential candidate must be enrolled in a cardiac rehabilitation program at screening or in the future.
  8. Implantable cardioverter defibrillator is required and must have been implanted a minimum of 30 days prior to screening.
  9. All male subjects regardless of fertility status or the fertility status of their partner must agree to use a condom and spermicide during any sexual relations for 6 months following IMP administration to protect their partner from potential viral shedding.
  10. All subjects regardless of fertility status or the fertility status of their partner must agree to have any male partner use a condom and spermicide during any sexual relations for 6 months following IMP administration to protect their partner from potential viral shedding.
  11. All subjects capable of procreation with their partners must agree to use adequate contraception for 6 months following IMP administration to avoid pregnancy (defined as oral or injectable contraceptives, intrauterine devices, surgical sterilization in addition to/or a combination of a condom and spermicide).
  12. Agree to not donate sperm or oocytes for 6 months following IMP administration.
  13. Ability to sign Informed Consent Form and Release of Medical Information Form.

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from the study:

  1. De novo diagnosis of heart failure.
  2. Any IV therapy with positive inotropes, vasodilators or diuretics within 30 days prior to screening or enrollment.
  3. Restrictive cardiomyopathy, obstructive cardiomyopathy, acute myocarditis, pericardial disease, amyloidosis, infiltrative cardiomyopathy, uncorrected thyroid disease or discrete left ventricular aneurysm.
  4. Cardiac surgery, percutaneous coronary intervention, valvuloplasty or valve replacement within 30 days prior to screening.
  5. Myocardial infarction (e.g., ST elevation myocardial infarction [STEMI] or large non-STEMI) within 90 days prior to screening. Large non-STEMI shall be defined >3x the upper limit of normal (ULN) for creatinine kinase test or >5x ULN for troponin.
  6. Prior heart transplantation, left ventricular reduction surgery (LVRS), cardiomyoplasty, passive restraint device (e.g., CorCap™ Cardiac Support Device), mechanical circulatory support device (MCSD) or cardiac shunt.
  7. Likely to receive cardiac resynchronization therapy, cardiomyoplasty, LVRS, conventional revascularization procedure or valvular repair in the 6 months following treatment.
  8. Likely need for an immediate heart transplant or MCSD implant due to hemodynamic instability.
  9. Prior coronary artery bypass graft(s) is not necessarily exclusionary. A potential candidate should be reviewed on a case-by-case basis by the treating interventionist, taking into account the dominance of the system, the accessibility of the graft(s) orifice, and the contribution of the graft vessel(s) and native coronary arteries to viable myocardial perfusion. The case and tentative infusion strategy must be discussed with the medical or safety officer prior to enrollment of the subject into the study.
  10. Known hypersensitivity to radiopaque agents used for angiography; history of or likely need for, high dose corticosteroid pretreatment prior to contrast angiography.
  11. Significant, in the opinion of the investigator, left main or ostial right coronary luminal stenosis.
  12. Liver function tests (alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase) >3x ULN, total bilirubin >2x ULN or known intrinsic liver disease (e.g., cirrhosis, chronic hepatitis B or hepatitis C virus infection).
  13. Current or likely need for hemodialysis within 12 months following enrollment or current glomerular filtration rate (GFR) ≤20 mL/minute/1.73 m^2 estimated by Modification of Diet in Renal Disease (MDRD) formula for calculating the GFR MDRD calculation.
  14. Bleeding diathesis or thrombocytopenia defined as platelet count <75,000 platelets/μL.
  15. Anemia defined as hemoglobin <9 g/dL.
  16. Diagnosis of, or treatment for, any cancer within the last 5 years except for basal cell carcinoma or carcinomas in situ where surgical excision was considered curative. (Past medical history of cancer is not exclusionary as long as the subject has been disease free for at least 5 years since the time of diagnosis and treatment).
  17. Previous participation in a study of gene transfer; however, if the study was unblinded or documentation otherwise exists that the subject was randomized to the placebo control group and did not receive active gene transfer agent, the subject may be considered for this study.
  18. Receiving investigational intervention or participating in another clinical study within 30 days or within 5 half-lives of the drug prior to screening. Exception may be made if the individual is enrolled in a non-therapeutic observational study (registry) or the observational portion of a therapeutic study where the sponsoring authority authorizes enrollment.
  19. Pregnancy or lactation.
  20. Recent history of psychiatric disease (including drug or alcohol abuse) that is likely to impair subject's ability to comply with protocol-mandated procedures, in the opinion of the investigator.
  21. Other concurrent medical condition(s) that, while not explicitly excluded by the protocol, could jeopardize the safety of the patient or objectives of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06-26 (Actual)

PRIMARY OUTCOMES:
Phase 1 and Phase 2: Safety profile of MYDICAR (proportion of subjects who complete the study; adverse event; concomitant medication use and changes in heart failure-related medications; incidence and event rates of hospitalizations | 24 months
  The primary objective of the study is to characterize the safety profile of MYDICAR. Safety outcomes will include proportion of subjects who complete the study; adverse event incidence, severity and relationship to investigational medicinal product or cardiac catheterization procedure; concomitant medication use and changes in heart failure-related medications; incidence and event rates of hospitalizations, ambulatory worsening of heart failure, myocardial infarction, stroke, mechanical circulatory support device (MCSD) implantation, heart transplant, and death; changes from baseline in laboratory tests, 12-lead electrocardiogram, and physical examination including weight and vital signs; and changes from baseline in implantable cardioverter defibrillator interrogation parameters.

OTHER OUTCOMES:
Phase 2: Rates of recurrent events (defined as hospitalizations for failure of the native heart that has not been implanted with an MCSD and/or ambulatory worsening failure of the native heart that has not been implanted with an MCSD) | 24 months
  Recurrent events are defined as hospitalizations for failure of the native heart that has not been implanted with an MCSD and/or ambulatory worsening failure of the native heart that has not been implanted with an MCSD.
Phase 2: Rates of terminal events (defined as all-cause death, MCSD implantation, or transplant) | 24 months
  Terminal events are defined as all-cause death, MCSD implantation, or transplant.
Phase 2: Change from baseline in left ventricular end systolic volume (LVESV) | 12 months
  Changes from baseline with positive values indicate a worsening in heart function and changes from baseline with negative values indicate an improvement in symptoms.
Phase 2: Change from baseline in distance walked during the 6-minute walk test (6MWT) | 12 months
  The 6MWT measures the distance walked in meters during a 6-minute test. Higher values indicate a better functional status. Changes from baseline with negative values indicate a worsening in function and changes from baseline with positive values indicate an improvement in function.
Phase 2: Change from baseline in Kansas City Cardiomyopathy Questionnaire [KCCQ] scores | 12 months
  The KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Phase 2: Change from baseline in New York Heart Association [NYHA] classification | 12 months
  NYHA classification is a symptomatic assessment in which the investigator evaluates subjects on a scale ranging from Class I (subjects with no limitation of activities, no symptoms from ordinary activities) to Class IV (subjects who should be at complete rest, confined to bed or chair; any physical activity brings on discomfort and symptoms occur at rest).
Phase 2: Change from baseline in N-terminal prohormone brain natriuretic peptide (NT-proBNP) levels | 12 months
  NT-proBNP is a biomarker for heart failure. Increased levels of this biomarker are associated with increased mortality and cardiovascular hospitalization in patients with heart failure.
Phase 1 and Phase 2: Transgene presence | 24 months
  The presence of AAV1/SERCA2a DNA will be evaluated by quantitative polymerase chain reaction (qPCR) in available tissue samples.
Phase 1 and Phase 2: SERCA2a expression | 24 months
  Gene expression of the SERCA2a transgene will be evaluated by reverse transcription qPCR in available tissue samples.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-858-366-4081, Study Director — Celladon Corporation
Locations (4):
- United States (4):
  - La Jolla, California
  - San Diego, California
  - Kansas City, Missouri
  - New York, New York

REFERENCES:
- [Background] Jaski BE, Jessup ML, Mancini DM, Cappola TP, Pauly DF, Greenberg B, Borow K, Dittrich H, Zsebo KM, Hajjar RJ; Calcium Up-Regulation by Percutaneous Administration of Gene Therapy In Cardiac Disease (CUPID) Trial Investigators. Calcium upregulation by percutaneous administration of gene therapy in cardiac disease (CUPID Trial), a first-in-human phase 1/2 clinical trial. J Card Fail. 2009 Apr;15(3):171-81. doi: 10.1016/j.cardfail.2009.01.013. PMID 19327618
- [Background] Jessup M, Greenberg B, Mancini D, Cappola T, Pauly DF, Jaski B, Yaroshinsky A, Zsebo KM, Dittrich H, Hajjar RJ; Calcium Upregulation by Percutaneous Administration of Gene Therapy in Cardiac Disease (CUPID) Investigators. Calcium Upregulation by Percutaneous Administration of Gene Therapy in Cardiac Disease (CUPID): a phase 2 trial of intracoronary gene therapy of sarcoplasmic reticulum Ca2+-ATPase in patients with advanced heart failure. Circulation. 2011 Jul 19;124(3):304-13. doi: 10.1161/CIRCULATIONAHA.111.022889. Epub 2011 Jun 27. PMID 21709064
- [Background] Zsebo K, Yaroshinsky A, Rudy JJ, Wagner K, Greenberg B, Jessup M, Hajjar RJ. Long-term effects of AAV1/SERCA2a gene transfer in patients with severe heart failure: analysis of recurrent cardiovascular events and mortality. Circ Res. 2014 Jan 3;114(1):101-8. doi: 10.1161/CIRCRESAHA.113.302421. Epub 2013 Sep 24. PMID 24065463